CLINICAL TRIAL: NCT05182957
Title: Clinical Study on the Efficacy and Safety of Anti-PD-1 Monoclonal Antibody Combined Lenalidomide and Azacitidine in Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Clinical Study on Anti-PD-1 Plus Lenalidomide and Azacitidine in Relapsed/Refractory Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/R PTCL 01
Record Dates: First submitted 2021-12-16; First posted 2022-01-10 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Relapsed/Refractory Peripheral T-cell Lymphoma
Keywords: Anti-PD-1 monoclonal antibody,Lenalidomide,Azacitidine
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — spartalizumab; Lenalidomide; Immunologic Factors; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 monoclonal antibody+Lenalidomide+Azacitidine (Experimental): Anti-PD-1 monoclonal antibody plus Lenalidomide, Azacitidine
  Interventions: Drug: Anti-PD-1 monoclonal antibody; Drug: Lenalidomide; Drug: Azacitidine

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — Anti-PD-1 monoclonal antibody, 200mg i.v d1 (/21d)
  Other Names: Anti-PD-1 antibody
Drug: Lenalidomide — Lenalidomide 25mg qd po d1-d10 (/21d)
  Other Names: Immunomodulator
Drug: Azacitidine — Azacitidine 75mg/m2 i.v d1-d7 (/21d)
  Other Names: 5-Ladakamycin

SUMMARY:
Aim of this study will evaluate the Efficacy and Safety of Anti-PD-1 monoclonal antibody Combined Lenalidomide and Azacitidine in Relapsed/Refractory Peripheral T-cell Lymphoma Patients.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCLs) are malignancies of immunologically mature T-cells that arise in peripheral lymphoid tissues. Compared with B-cell lymphoma, the treatment methods of PTCL are more limited, the first-line therapy is usually CHOP-like therapy, but the efficacy is poor, 5-year overall survival rate (OS) is only 30%-40%. Anti-PD-1 monoclonal antibody, Lenalidomide and Azacitidine can all have tumor-killing effects, and the three have complementary theoretical basis in the mechanism of action. This study will evaluate the efficacy and safety of Anti-PD-1 monoclonal antibody Combined Lenalidomide and Azacitidine in Relapsed/Refractory Peripheral T-cell Lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological immunohistochemistry or flow cytometry confirmed that R/R PTCL with measurable (diameter greater than 1.5cm) lesions meets any of the following conditions: 1> After 4 courses of standard first-line therapy or 2 courses of more than two-line therapy, the lesions were reduced by <50%; 2> PTCL with disease progression after first-line or induction therapy; 3> After hematopoietic stem cell transplantation, new lesions appear or the size of previously affected lesions increased by more than 50%.
2. Age ≥ 18 years.
3. ECOG≤2分.
4. The main organ functions need to meet the following conditions:Hemogram needs to meet HB ≥70*1012/L，PLT≥50*109/L，NE≥1*109/L；LVEF≥50%;CR≤132umol/l or CCr≥60 ml/min;ALT and AST≤2 times normal range；Lung function≤Level 1;dyspnea(CTCAE v5.0),and blood oxygen saturation without oxygen absorption> 91%.
5. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study until the follow-up one year period of the study.
6. Estimated survival time ≥3 months.
7. Voluntary signing of informed consent.

Exclusion Criteria:

1. Accepted major surgery within 4 weeks before treatment.
2. Prior malignancy (other than Relapsed/Refractory Peripheral T-cell Lymphoma), except for cured malignant tumors with no active lesions for 3 years;Adequate treatment of inactive lesions in non-melanoma skin cancer,malignant tonsilloma or carcinoma in situ;
3. Patients who have previously received failed allogeneic hematopoietic stem cell transplantation.
4. Have stroke or intracranial hemorrhage within 3 months.
5. Evidence of complications or medical conditions, including but not limited, that may interfere the conduct of the study or place the patient at serious risk:significant cardiovascular disease(class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification、myocardial infarction within 6 months of screening、uncontrolled or symptomatic arrhythmias) and/or significant lung disease.
6. HIV infection and/or active hepatitis B or active hepatitis C.
7. Uncontrolled systemic infection.
8. Pregnant or breasting-feeding women.
9. According to the researchers' judgment, any life-threatening disease, medical condition or organ system dysfunction which can endanger the patient's safety and Interfer with the absorption or metabolism of anti-PD-1 monoclonal antibody plus Lenalidomide and Azacitidine,may put the results of a study at unnecessary risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-12-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | up to 12 months
  To measure the duration of response to Anti-PD-1 antibody plus Lenalidomide and Azacitidine over a follow-up period of 12 months
Overall Response Rate (ORR) | up to 12 months
  To measure the duration of response to Anti-PD-1 antibody plus Lenalidomide and Azacitidine over a follow-up period of 12 months

SECONDARY OUTCOMES:
Complete Response Rate | up to 12 months
  Number of patients who achieved complete response after treatment by Anti-PD-1 antibody plus Lenalidomide and Azacitidine
Duration of Response | up to 12 months
  Duration of overall response will be assessed from the first Anti-PD-1 antibody plus Lenalidomide and Azacitidine given to progression,death or last follow-up.
Overall Survival | up to 12 months
  OS will be assessed from the first Anti-PD-1 antibody plus Lenalidomide and Azacitidine given to death or last follow-up.
Adverse events profile | Measured from start of treatment until 28 days after last dose
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China